CLINICAL TRIAL: NCT00577252
Title: Coping Compliance and Adjustment in Adolescents With Cystic Fibrosis
Status: Completed | Type: Observational
Sponsor: Akron Children's Hospital (Other)
Responsible Party: Nathan Kraynack, MD, Akron Children's Hospital
Other Study IDs: COPING1424; COPING1424
Record Dates: First submitted 2007-12-18; First posted 2007-12-20 (Estimated); Last update posted 2009-11-24 (Estimated); Status verified 2009-11

CONDITIONS: Cystic Fibrosis
Keywords: Cystic fibrosis; Adolescents; Coping Compliance; Adjustment
MeSH Terms: conditions — Cystic Fibrosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- 1: Adolescents with CF.

SUMMARY:
In this research, we will use established surveys to look at the relationship between various styles of coping with a disease, religious coping styles, treatment compliance, locus of control, broad measures of mental health and adjustment, and basic health data (e.g., PFTs, recent hospitalizations or antibiotics within the past year, lung microbiology, CFTR mutations, and co-morbid conditions such as diabetes, depression, and liver disease). While the research is correlational, it should suggest relationships (both positive and negative) between various coping styles and desired outcomes (compliance and well-being).

DETAILED DESCRIPTION:
OVERVIEW: We anticipate that the data we collect will help us better understand some of the factors associated with improved coping, treatment compliance, and emotional adjustment, which, in turn, may suggest possible interventions to improve compliance, emotional adjustment, and general physical health. Specific hypotheses include the following:

1. Subjects who score high on measures of positive coping will have greater levels of treatment compliance and psychological well-being.
2. Subjects who score high on measures of negative coping will have lower levels of treatment compliance and psychological well-being.
3. Subjects who score high on measures of positive religious coping will have greater levels of treatment compliance and psychological well being.
4. Subjects who score high on measures of negative religious coping will have lower levels of treatment compliance and psychological well-being.
5. Subjects who score high on measures of internal locus of control will have higher levels of treatment compliance and psychological well-being compared to subjects who score low on measures of internal locus of control.
6. Subjects who score high on measures of treatment compliance will have higher levels of physical health.
7. We do not anticipate a positive correlation between positive coping mechanisms and general physical health; however, subjects who score high on measures of negative coping may have lower levels of general physical health (e.g., lower PFTs, increased rates and lengths of hospitalizations) probably due to third variables (e.g., if someone uses denial as a coping mechanism, it may lead to poor treatment compliance, which may lead to declines in physical health).
8. Anecdotal evidence suggests that parental education may be positively correlated with treatment compliance, but this has not been evaluated. Likewise, anecdotal evidence suggest that marital status may be correlated with treatment compliance (probably because of third variables, e.g., if, as much research suggests, divorce is related to lower SES and fewer social supports, these factors may in turn interfere with treatment compliance). Two questions on the demographic sheet will allow us to explore whether or not this may be worth exploring further.

ELIGIBILITY:
Inclusion Criteria:

* cystic fibrosis age 13-19 yrs

Exclusion Criteria:

* acutely ill

Ages: 13 Years to 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Adolescents age 13-19 with CF at a single CF center.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2007-10; Study Completion 2008-04 (Actual)

PRIMARY OUTCOMES:
Multiple measures of coping strategies in adolescents with cystic fibrosis. | Single visit

SECONDARY OUTCOMES:
Coping startegies will be correlated with measures of clinical illness. | Single visit

CONTACTS AND LOCATIONS:
Overall Officials: Nathan C Kraynack, MD, Principal Investigator — Akron Children's Hospital
Locations (1):
- Akron Children's Hospital, Akron, Ohio, United States